CLINICAL TRIAL: NCT07334405
Title: Prospective Study on Therapeutic Approaches in Dental Traumatology: Management of Traumatic Tooth Avulsion
Brief Title: Dental Trauma - Avulsion
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Antonio Barone, Full Professor, University of Pisa
Other Study IDs: Dental Trauma - Tooth avulsion
Record Dates: First submitted 2025-12-18; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Dental Trauma
Keywords: trauma; avulsion; permanent tooth
MeSH Terms: conditions — Wounds and Injuries; Fractures, Avulsion | interventions — Tooth Replantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dental avulsion: Adult and pediatric patients who experienced a traumatic avulsion of one or more permanent teeth
  Interventions: Other: Tooth replantation

INTERVENTIONS:
Other: Tooth replantation — Avulsed teeth were replanted according to the International Academy of Dental Traumatology guidelines (IADT)

SUMMARY:
Dental traumatology is a field of dentistry , especially in pediatric age, but also in adulthood with permanent dentition. Dental trauma has a higher incidence in preschool, school-age, and adolescent patients, accounting for about 5% of injuries for which the intervention of a specialist physician is required. Traumatic avulsion of permanent teeth accounts up to 0.5-16% of all dental injuries and is considered one of the true emergencies in dentistry.The treatment of choice in case of traumatic avulsion of permanent teeth is the quickest-as-possible replantation. The primary objectives of this prospective study were to evaluate the incidence of complications and survival rates of replanted teeth over time. The secondary objectives were to assess and to examine the correlation between the development of complications and factors such as extra-oral time, storage media, root maturity and the presence of alveolar fractures.

ELIGIBILITY:
Inclusion criteria

* Adult and pediatric patients who experienced a dental trauma
* Adult and pediatric patients who experienced a traumatic avulsion of one or more permanent teeth
* Patients treated with dental replantation following the International Association of Dental Traumatology (IADT) guidelines
* Availability of clinical and radiographic follow-up for at least one year

Exclusion criteria

- Patients with absolute contraindications to dental replantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult and pediatric patients who experienced a traumatic avulsion of one or more permanent teeth and were treated at the University Hospital of Pisa
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2031-11-20 (Estimated)

PRIMARY OUTCOMES:
Tooth survival | 2 weeks after trauma
  Tooth survival was defined as the presence of the tooth in the oral cavity at the time of follow-up. Tooth survival is assessed at each follow-up visit after replantation following IADT guidelines.
Tooth survival | 4 weeks after trauma
  Tooth survival was defined as the presence of the tooth in the oral cavity at the time of follow-up. Tooth survival is assessed at each follow-up visit after replantation following the IADT guidelines.
Tooth survival | 3 months after trauma
  Tooth survival was defined as the presence of the tooth in the oral cavity at the time of follow-up. Tooth survival is assessed at each follow-up visit after replantation following the IADT guidelines.
Tooth survival | 6 months after trauma
  Tooth survival was defined as the presence of the tooth in the oral cavity at the time of follow-up. Tooth survival is assessed at each follow-up visit after replantation following the IADT guidelines.
Tooth survival | 12 months after trauma
  Tooth survival was defined as the presence of the tooth in the oral cavity at the time of follow-up. Tooth survival is assessed at each follow-up visit after replantation following the IADT guidelines.
Tooth survival | 24 months after trauma
  Tooth survival was defined as the presence of the tooth in the oral cavity at the time of follow-up. Tooth survival is assessed at each follow-up visit after replantation following the IADT guidelines.
Tooth survival | 36 months after trauma
  Tooth survival was defined as the presence of the tooth in the oral cavity at the time of follow-up. Tooth survival is assessed at each follow-up visit after replantation following the IADT guidelines.
Tooth survival | 48 months after trauma
  Tooth survival was defined as the presence of the tooth in the oral cavity at the time of follow-up. Tooth survival is assessed at each follow-up visit after replantation following the IADT guidelines.
Tooth survival | 60 months after trauma
  Tooth survival was defined as the presence of the tooth in the oral cavity at the time of follow-up. Tooth survival is assessed at each follow-up visit after replantation following the IADT guidelines.
Incidence of complications | 2 weeks after trauma
  Evaluated as presence/absence of a dental complication following trauma.
Incidence of complications | 4 weeks after trauma
  Evaluated as presence/absence of a dental complication following trauma.
Incidence of complications | 3 months after trauma
  Evaluated as presence/absence of a dental complication following trauma.
Incidence of complications | 6 months after trauma
  Evaluated as presence/absence of a dental complication following trauma.
Incidence of complications | 12 months after trauma
  Evaluated as presence/absence of a dental complication following trauma.
Incidence of complications | 24 months after trauma
  Evaluated as presence/absence of a dental complication following trauma.
Incidence of complications | 36 months after trauma
  Evaluated as presence/absence of a dental complication following trauma.
Incidence of complications | 48 months after trauma
  Evaluated as presence/absence of a dental complication following trauma.
Incidence of complications | 60 months after trauma
  Evaluated as presence/absence of a dental complication following trauma.

SECONDARY OUTCOMES:
Dental mobility | 2 weeks after trauma
  Tooth mobility clinically evaluated from 0 to 3
Dental mobility | 4 weeks after trauma
  Tooth mobility clinically evaluated from 0 to 3
Dental mobility | 3 months after trauma
  Tooth mobility clinically evaluated from 0 to 3
Dental mobility | 6 months after trauma
  Tooth mobility clinically evaluated from 0 to 3
Dental mobility | 12 months after trauma
  Tooth mobility clinically evaluated from 0 to 3
Dental mobility | 24 months after trauma
  Tooth mobility clinically evaluated from 0 to 3
Dental mobility | 36 months after trauma
  Tooth mobility clinically evaluated from 0 to 3
Dental mobility | 48 months after trauma
  Tooth mobility clinically evaluated from 0 to 3
Dental mobility | 60 months after trauma
  Tooth mobility clinically evaluated from 0 to 3
Complication - root resorption | 2 weeks after trauma
  Radiographic signs of root resorption
Complication - root resorption | 4 weeks after trauma
  Radiographic signs of root resorption
Complication - root resorption | 3 months after trauma
  Radiographic signs of root resorption
Complication - root resorption | 6 months after trauma
  Radiographic signs of root resorption
Complication - root resorption | 12 months after trauma
  Radiographic signs of root resorption
Complication - root resorption | 24 months after trauma
  Radiographic signs of root resorption
Complication - root resorption | 36 months after trauma
  Radiographic signs of root resorption
Complication - root resorption | 48 months after trauma
  Radiographic signs of root resorption
Complication - root resorption | 60 months after trauma
  Radiographic signs of root resorption
Complication - ankylosis | 2 weeks after trauma
  Clinical and radiographic signs of ankylosis (loss of periodontal space, absence of physiological tooth mobility)
Complication - ankylosis | 4 weeks after trauma
  Clinical and radiographic signs of ankylosis (loss of periodontal space, absence of physiological tooth mobility)
Complication - ankylosis | 3 months after trauma
  Clinical and radiographic signs of ankylosis (loss of periodontal space, absence of physiological tooth mobility)
Complication - ankylosis | 6 months after trauma
  Clinical and radiographic signs of ankylosis (loss of periodontal space, absence of physiological tooth mobility)
Complication - ankylosis | 12 months after trauma
  Clinical and radiographic signs of ankylosis (loss of periodontal space, absence of physiological tooth mobility)
Complication - ankylosis | 24 months after trauma
  Clinical and radiographic signs of ankylosis (loss of periodontal space, absence of physiological tooth mobility)
Complication - ankylosis | 36 months after trauma
  Clinical and radiographic signs of ankylosis (loss of periodontal space, absence of physiological tooth mobility)
Complication - ankylosis | 48 months after trauma
  Clinical and radiographic signs of ankylosis (loss of periodontal space, absence of physiological tooth mobility)
Complication - ankylosis | 60 months after trauma
  Clinical and radiographic signs of ankylosis (loss of periodontal space, absence of physiological tooth mobility)
Extra-oral time | At baseline (toorh replantation after avulsion)
  Evaluated in minutes from the avulsion to the replantation
Storage medium | At baseline (tooth replantation following avulsion)
  Storage medium of the avulsed tooth (milk, water, saline, etc)
Alveolar fracture | At baseline (tooth replantation following avulsion)
  Presence of alveolar fractures associated to tooth avulsion

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Pisa, Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No